CLINICAL TRIAL: NCT04143386
Title: Prognostic Hemodynamic and Metabolic Profiles of Late Stage Lower Extremity Arterial Disease
Acronym: PREDICTOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Tartu (Other)
Collaborators: Estonian Science Foundation (Other Government); Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Jaak Kals, Principal Investigator, University of Tartu
Other Study IDs: 283T10
Record Dates: First submitted 2019-10-24; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Lower Extremity Arterial Disease (Fontaine Stages IIb-IV)
Keywords: lower extremity arterial disease; hemodynamics; arterial stiffness; metabolism; metabolomics; inflammation; oxidative stress; biomarkers; prognosis
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Late stage lower extremity arterial disease (LEAD) is known to be associated with hemodynamic and metabolic abnormalities and very poor long-term prognosis. The prognostic value of hemodynamic and metabolic profiling, however, is yet to be determined in this patient group.

Current study aims to identify novel prognostic biomarkers for better risk stratification of late stage LEAD patients. It also allows to determine associations between hemodynamic/arterial stiffness indices, low-molecular weight metabolites and other substances (e.g. mediators of inflammation and bone-mineral metabolism, cardiac and kidney injury biomarkers, microRNAs) thus providing potentially valuable insight into the pathogenic mechanisms of this disease.

ELIGIBILITY:
Exclusion Criteria:

* Fontaine stage I-IIa;
* acute limb ischemia;
* age <35 or >85 years;
* fasting < 6 hours;
* time since the last use of tobacco products < 4 hours;
* body mass index ≥ 40 kg/m2
* blood pressure ≥ 180/120mmHg;
* unstable angina;
* atrial fibrillation at the time of presentation;
* myocardial infarction, stroke or TIA during the preceding 3 months;
* any revascularization during the preceding 1 month;
* severe heart failure (NYHA IV);
* clinically significant heart valve disease;
* severe physical disability (other than limb ischemia);
* acute infectious disease;
* active malignancy or chemotherapy or disease-free < 5 years;
* type 1 diabetes;
* uncompensated thyrotoxicosis/hypothyroidism or other clinically significant endocrine disorders;
* moderate to severe asthma (GINA 2016);
* severe chronic obstructive pulmonary disease (mMRC grade 3-4)
* acute (KDIGO 2012) or chronic renal disease (eGFR-EPI <30mL/min/1.73 m2);
* clinically significant acute or chronic liver disease;
* severe anemia (<80 g/L);
* clinically significant neuroinflammatory or neurodegenerative disease;
* active rheumatism;
* clinically significant connective tissue disease;
* alcoholism or drug abuse;
* psychotic disorders

Ages: 35 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic lower extremity arterial disease referred to Tartu University Hospital for revascularization (angioplasty/stenting or bypass surgery).
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2019-11-04 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of major adverse cardiovascular events, major adverse limb events and deaths | 5 years
  A composite of any of the following events, as documented by patients' hospital or death records:
  1. nonfatal myocardial infarction or stroke
  2. fatal myocardial infarction or stroke
  3. hospitalization for angioplasty or bypass surgery for coronary or peripheral vessel disease
  4. LEAD-related major lower extremity amputation
  5. other cardiovascular deaths (cardiac arrest, lethal arrhythmia, heart failure, aortic dissection or rupture)
  6. non-cardiovascular deaths

SECONDARY OUTCOMES:
Number of fatal cardiovascular events | 5 years
Number of non-fatal cardiovascular events | 5 years
Number of LEAD-related major lower extremity amputations | 5 years
Number of hospitalizations for angioplasty or bypass surgery for coronary or peripheral vessel disease | 5 years
Number of deaths from all causes | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jaak Kals, MD, PhD, Principal Investigator — University of Tartu; Jaan Eha, MD, PhD, Study Chair — University of Tartu; Mihkel Zilmer, dr. med., Study Chair — University of Tartu; Kaido Paapstel, MD, PhD, Study Director — University of Tartu; Kaspar Tootsi, MD, PhD, Study Chair — University of Tartu; Karl Kuusik, MD, Study Chair — University of Tartu; Tuljo Ööbik, MD, Study Chair — University of Tartu; Riina Kaur, Study Chair — University of Tartu
Locations (1):
- Tartu University Hospital, Tartu, Tartu, Estonia

REFERENCES:
- See also: Endothelial Research Centre — https://endothelialcentre.ut.ee/